CLINICAL TRIAL: NCT00695227
Title: Screening for Barrett's Esophagus in Otolaryngology Patients
Acronym: SCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K23 DK66165 (completed); K23DK066165 (NIH)
Record Dates: First submitted 2008-06-06; First posted 2008-06-11 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Extraesophageal Symptoms; Cough; Throat Clearing; Hoarseness; Difficulty Swallowing
Keywords: laryngopharyngeal reflux; extraesophageal reflux symptoms
MeSH Terms: conditions — Cough; Hoarseness; Deglutition Disorders; Laryngopharyngeal Reflux | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening for Barrett's Esophagus (Experimental)
  Interventions: Diagnostic Test: Screening for Barrett's Esophagus

INTERVENTIONS:
Diagnostic Test: Screening for Barrett's Esophagus

SUMMARY:
The purpose of this project is to develop an accurate method to identify patients that suffer from acid reflux, but may not present with classic reflux symptoms (such as heart burn). Additionally, it is the purpose of this project to utilize the Unsedated Small-caliber Endoscopy (USE) to assess the prevalence of Barrett's esophagus in a population of patients with laryngopharyngeal reflux (LPR) symptoms and to define normal patterns of LPR. Laryngopharyngeal reflux (LPR) is when a small amount of stomach contents and acid are pushed up through the esophagus and may affect the vocal cords and upper respiratory tract.

It is suspected that patients with LPR symptoms may have a prevalence of Barrett's esophagus similar to that found in a population with typical reflux symptoms. We propose to systematically test this hypothesis using the USE.

This project is designed to improve the methods of identifying patients with a form of acid reflux that is often undetected, and thus untreated. If this project is successful then more patients with Barrett's esophagus will be identified; furthermore, screening and treatment for this pre-cancerous condition will be improved.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Prior anti-reflux surgery, laryngeal surgery, trauma to larynx Esophageal diverticulum Pregnancy Anticoagulation therapy Esophageal varices ENT malignancy History of recurrent epistaxis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary aim of the study is to establish that patients with symptoms of LPR who are referred to an otolaryngology clinic have a prevalence of Barrett's metaplasia equivalent to that of a population with GERD symptoms. | One time

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Schindler, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Nason KS, Murphy T, Schindler J, Schipper PH, Hoppo T, Diggs BS, Sauer DA, Shaheen NJ, Morris CD, Jobe BA; Barrett's Esophagus Risk Consortium (BERC). A cross-sectional analysis of the prevalence of Barrett esophagus in otolaryngology patients with laryngeal symptoms. J Clin Gastroenterol. 2013 Oct;47(9):762-8. doi: 10.1097/MCG.0b013e318293d522. PMID 23751847